CLINICAL TRIAL: NCT06158490
Title: An Efficacy and Safety Study of JYP0061 Tablets in Adult Patients With Moderate-to-Severe Atopic Dermatitis: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2 Clinical Trial
Brief Title: A Study to Evaluate JYP0061 Tablets in Patients With Moderate-to-severe Atopic Dermatitis
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou JOYO Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JYP0061M210
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-11

CONDITIONS: Moderate-to-severe Atopic Dermatitis
Keywords: atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JYP0061 15 mg Group (Experimental): Participants in this arm will receive 15 mg of JYP0061 once daily for a total treatment period of 12 weeks.
  Interventions: Drug: JYP0061 15 mg
- JYP0061 30 mg Group (Experimental): articipants in this arm will receive 30 mg of JYP0061 once daily for a total treatment period of 12 weeks.
  Interventions: Drug: JYP0061 30 mg
- Placebo Group (Placebo Comparator): Participants in this arm will receive a placebo once daily for a total treatment period of 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JYP0061 15 mg — Participants in the JYP0061 15 mg group will receive a 15 mg oral tablet of JYP0061 once daily for 12 weeks.
  Arms: JYP0061 15 mg Group
Drug: JYP0061 30 mg — articipants in the JYP0061 30 mg group will receive a 30 mg oral tablet of JYP0061 once daily for 12 weeks.
  Arms: JYP0061 30 mg Group
Drug: Placebo — Participants in the placebo group will receive a matching placebo tablet once daily for 12 weeks.
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of JYP0061 in adult patients with moderate-to-severe atopic dermatitis. The main questions it aims to answer are:

* The efficacy of JYP0061 in treating adult patients with moderate-to-severe atopic dermatitis.
* The safety profile of JYP0061 when administered to adult patients with moderate-to-severe atopic dermatitis.

Participants will:

* Be treated with either a low-dose or high-dose of JYP0061.
* Undergo efficacy and safety evaluations as stipulated in the trial protocol.

DETAILED DESCRIPTION:
The goal of this clinical trial is to assess JYP0061 for efficacy and safety in adult patients with moderate-to-severe atopic dermatitis. The main objectives it aims to address are the determination of the drug's therapeutic effect and its safety profile in this patient population. Upon providing written informed consent after being briefed on the study details and potential risks, participants will enter a screening period of up to 4 weeks to confirm their eligibility.

The main tasks for participants will include:

* Being randomized to receive either a low-dose or high-dose of JYP0061.
* Completing a treatment course of 12 weeks.
* Undergoing efficacy and safety assessments as prescribed by the study's protocol.

Following the treatment phase, all participants, whether they have completed the treatment course on schedule or have discontinued early, will be monitored for an additional 4 weeks to further evaluate safety post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* The age of the participants should be between 18 and 65 years old, with no restrictions on gender.
* Participants must weigh 40 kg or more
* At the time of screening, participants must meet the Williams criteria for atopic dermatitis, have had the condition for at least one year, and the severity of the disease should be moderate to severe;
* Participants agree from the time of signing the informed consent form until the completion of the study's final visit to use only non-medicated emollients (moisturizing creams) or other concomitant treatments allowed by the protocol.
* Fully understand the purpose and requirements of this trial, voluntarily participate, and sign the written informed consent form, and are able to complete the study according to its requirements.

Exclusion Criteria:

* Suspected or confirmed allergy to any component of the study drug or similar ingredients, or having a history of moderate allergic diseases (such as food allergies, drug allergies, etc., except for allergies related to atopic dermatitis) at the time of signing the informed consent form;
* At the time of screening, having other skin diseases or skin infections that could affect the evaluation of the trial results, or having extensive tattoos, birthmarks, skin scars, etc., in the area of skin lesions, aside from atopic dermatitis;
* Having or having had other connective tissue diseases, apart from a history of atopic dermatitis;
* Participation in another clinical trial within one month prior to screening or within five half-lives of the investigational drug (whichever is longer);
* Underwent major surgery within 12 weeks prior to screening;
* Conditions that negatively affect the immune response (such as history of organ transplantation), or subjects with known immunodeficiency syndromes (acquired immunodeficiency syndrome, genetic immunodeficiency, and drug-induced immunodeficiency).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving at least a 75% reduction in Eczema Area and Severity Index (EASI 75) from baseline. | Evaluations will be conducted weekly for up to 12 weeks
  The Eczema Area and Severity Index (EASI) is a measure of eczema severity, combining area coverage and symptom intensity (erythema, edema/papulation, excoriation, lichenification) for four body regions. EASI scores range from 0 (no eczema) to 72 (maximum severity), with higher scores indicating worse outcomes. This primary outcome assesses the proportion of participants who achieve at least a 75% reduction in EASI from baseline to Week 12.

SECONDARY OUTCOMES:
Proportion of participants achieving EASI 75 at Weeks 2, 4, and 8. | Weeks 2, 4, and 8.
  Percentage of participants achieving a 75% reduction in EASI from baseline at each specified week.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China